CLINICAL TRIAL: NCT04918849
Title: Characterising the Spread of COVID-19 Misinformation Through WhatsApp in India
Brief Title: WhatsApp in India During the COVID-19 Pandemic
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yale-NUS College (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-CERC-001C
Record Dates: First submitted 2021-06-08; First posted 2021-06-09 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-06

CONDITIONS: Covid19
Keywords: WhatsApp; Misinformation; Rumours; India; Experience Sampling
MeSH Terms: conditions — COVID-19; Communication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Community Sample: We plan to recruit a community sample of 1000 from the Indian Population.

SUMMARY:
Digital misinformation has been flagged as a major risk of the 21st century, with an estimated cost of $78 billion to the global economy each year. Given this scope, we propose to characterize how misinformation is spread via messenger platforms (e.g. WhatsApp).

Specifically, we seek to:

1. Identify metrics of potential misinformation (Aim 1). This is based on the hypothesis that although message contents are highly private, proxy markers can be used to identify potential misinformation.
2. Understand the base-rate by which misinformation is shared via messaging applications (Aim 2). This is founded on the hypothesis that misinformation is endemic on messaging platforms, and thus needs to be documented.
3. Identify "super spreaders" responsible for sending and receiving a large volume of misinformation (Aim 3). Here, we hypothesise that a small group of super spreaders are responsible for the bulk of misinformation-sharing on messaging applications.

The thrust of this work aligns with both government priorities and the grant's thematic areas, providing actionable findings that are timely amidst a worldwide surge of misinformation.

ELIGIBILITY:
Inclusion Criteria:

* Lived in India for more than 2 years,
* Currently Living in India
* Owns a WhatsApp account

Exclusion Criteria:

* Not currently living in India
* Below the ages of 21
* Has not lived in India for more than 2 years
* does not own a WhatsApp account
* Does not speak English or Hindi

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A community sample of the 1000 people from the Indian population
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-05-21 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
WhatsApp Usage | 1 week, starting from date after baseline survey completion
  Participants were asked a series of questions daily related to their WhatsApp usage behaviors - in particular, their message-forwarding, personal chat and group chat behaviors.
Changes in fear with regards the COVID-19 situation across 1 week | 1 week, starting from date after baseline survey completion
  1 item each day on fear specifically of the COVID-19 situation (measured on a 4 point scale: min = 1, max = 4; higher scores indicating greater fear about the outbreak).
Changes in amount of thinking about the COVID-19 situation across 1 week | 1 week, starting from date after baseline survey completion
  1 item each day on how much they thought about the outbreak that day (measured on a 5 point scale: min = 1, max = 5; higher scores indicating more thinking about the outbreak).

CONTACTS AND LOCATIONS:
Locations (1):
- Yale-NUS College, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
Due to stipulations by the institutional review board, data can not be shared